CLINICAL TRIAL: NCT01622166
Title: Art Therapy for Symptom Reduction in Acute Schizophrenia - a Randomised Controlled Trial (Kunsttherapie Zur Symptomreduktion Bei Akuter Schizophrenie - Eine Randomisierte Kontrollierte Pilotstudie)
Brief Title: Art Therapy in Acute Schizophrenia
Acronym: KUSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Prof. K. Dannecker, Kunsttherapie Berlin Kunsthochschule Berlin-Weißensee (Unknown)
Responsible Party: Principal Investigator, Christiane Montag MD, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA1/104/11
Record Dates: First submitted 2012-06-12; First posted 2012-06-19 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- art therapy (Experimental): 12 sessions of art therapy / 6 weeks
  Interventions: Behavioral: psychodynamic art therapy
- TAU (No Intervention): treatment as usual / 6 weeks

INTERVENTIONS:
Behavioral: psychodynamic art therapy — 2 sessions à 1.5 hrs /week, intervention duration 6 weeks
  Arms: art therapy

SUMMARY:
Randomised, controlled, single-blinded pilot study to assess the efficacy of psychodynamic art therapy in a sample of hospitalized, (sub)acutely psychotic patients with a diagnosis of schizophrenia compared to a group of patients receiving treatment as usual.

*Main hypothesis: Art therapy has no impact on clinical symptoms and the course of remission compared to TAU.

*Exploratory hypotheses: Art therapy has no influence on quality of life, mentalizing function, self-efficacy and neuroleptic dosage compared to TAU.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia according to DSM-IV-TR
* age 18-64 yrs
* sufficient German language competency
* written informed consent

Exclusion Criteria:

* axis-I mental disorders other than schizophrenia
* comorbid antisocial personality disorder, relevant substance abuse,
* relevant severe somatic disease
* acute suicidal tendencies or aggression
* incapability to tolerate group settings

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Syndrome Scale (PANSS-) scores | weeks 0, 6, 12
  assessment of change of schizophrenic positive, negative and general symptom scores
safety measures | weeks 0, 6, 12
  number of participants with adverse events
Change in Calgary depression Scale (CDS-) scores | weeks 0, 6, 12
  assessment of change of depressive symptoms in schizophrenic patients as reflected by CDS-scores

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Montag, M.D., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Psychiatrische Universitätsklinik der Charité im St. Hedwig Krankenhaus, Berlin, Germany

REFERENCES:
- [Derived] Montag C, Haase L, Seidel D, Bayerl M, Gallinat J, Herrmann U, Dannecker K. A pilot RCT of psychodynamic group art therapy for patients in acute psychotic episodes: feasibility, impact on symptoms and mentalising capacity. PLoS One. 2014 Nov 13;9(11):e112348. doi: 10.1371/journal.pone.0112348. eCollection 2014. PMID 25393414
- See also: Related Info — http://www.kunsttherapie-berlin.de/